CLINICAL TRIAL: NCT01991964
Title: The Yield of Laryngeal Ultrasound in the Diagnosis of Laryngomalacia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TASMC-13-FS-0563-13-CTIL
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Stridor; Laryngomalacia
Keywords: stridor; laryngomalacia; ultrasound
MeSH Terms: conditions — Respiratory Sounds; Laryngomalacia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- laryngeal ultrasound stridor (Experimental): During the study period, infants referred for FLB and bronchoscopy due to congenital stridor at the Department of Pediatric Pulmonology, Critical Care and Sleep Medicine at the Tel Aviv Sourasky Medical Centre will undergo an awake US of the larynx prior to performing the Flexible bronchoscopy.
  Interventions: Other: laryngeal ultrasound
- laryngeal ultrasound -control (Other): Infants matched for age referred for flexible bronchoscopy for reasons other than stridor will undergo an awake US of the larynx.
  Interventions: Other: laryngeal ultrasound

INTERVENTIONS:
Other: laryngeal ultrasound

SUMMARY:
The hypothesis of the study is that laryngeal US can accurately and reliably diagnose laryngomalacia in infants with congenital stridor.

Stridor is a respiratory noise caused by partial obstruction of the large airways at the level of the pharynx, larynx and/or trachea. The most prevalent congenital cause of stridor is laryngomalacia. Flexible laryngobronchoscopy (FLB) under sedation is regarded as the gold standard. However, FLB under sedation has some drawbacks as it requires venous access, use of sedative agents, may cause discomfort for the patient and is costly.

Ultrasound (US) is a noninvasive, painless, radiation free, well tolerated imaging technique. It allows for dynamic assessment of moving structures in an awake patient and the results can be easily displayed and recorded.

ELIGIBILITY:
Inclusion Criteria:

Infants referred for FLB and bronchoscopy due to congenital stridor at the Department of Pediatric Pulmonology, Critical Care and Sleep Medicine at the Tel Aviv Sourasky Medical Centre

Exclusion Criteria:

* Prior knowledge of the cause for stridor
* History of foreign body aspiration

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The yield of US in diagnosing laryngomalacia in comparison to FLB. | December 2013- January 2015 (13 months)

SECONDARY OUTCOMES:
The yield of US in diagnosing other causes of congenital stridor compared to FLB. | December 2013- January 2015 (13 months)